CLINICAL TRIAL: NCT00844363
Title: Mechanism of Action of Narrowband UVB Phototherapy in the Treatment of Psoriasis Vulgaris
Brief Title: Narrowband UVB Phototherapy in the Treatment of Psoriasis Vulgaris
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to isolate sufficient cells from the skin biopsy to perform study related experiments
Sponsor: Rockefeller University (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Michelle Lowes, Rockefeller University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLO-0651
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NB-UVB (Other): Regular, monitored NB-UVB treatment. Patients will be treated 3 times per week, and a full course of therapy is 12 weeks. NB-UVB dosing is increased by 5-20% increments in exposure time, depending on response of the patient.
  Interventions: Procedure: NB-UVB

INTERVENTIONS:
Procedure: NB-UVB — UVB light will be administered to the entire body except for the genitals in men and eyelids, which will be shielded.NB-UVB dosing is increased by 5-20% increments in exposure time, depending on response of the patient.
  Other Names: narrowband UVB phototherapy

SUMMARY:
Ultra-violet light B (UVB) therapy has been used by dermatologists to treat psoriasis for decades. Only a few studies have begun to dissect the mechanism of how NB-UVB therapy causes lesion resolution. Results from this study will aid in identifying other diseases that may be treated successfully with NB-UVB. If we can identify the mechanism of action of this therapy, this may give us additional new therapeutic targets for psoriasis and other diseases. Our overall hypothesis is that UVB induces changes that will indicate a mechanism of action of this therapy in psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* History of chronic plaque psoriasis vulgaris, for at least six months.
* ≥10% body surface affected
* Age 18 or greater.
* Concomitant, chronic, but well-controlled medical conditions such as hypertension are allowable.
* No treatment with topical steroids for at least 2 weeks prior to entering the study
* No treatment with systemic therapies, including etretinate, UVB, PUVA, or cyclosporine, other biologics 4 weeks prior to entering the study. However, if a patient is considered to be "unstable", or would deteriorate clinically if the systemic agent is ceased (eg efalizumab), a shorter "washout" period may be considered, and would be documented in the patient charts.
* Patients who receive a stable dose of methotrexate (defined as <15mg/week for 4 months or greater) for psoriatic arthritis may be included.

Exclusion Criteria:

* Subjects who do not meet the above criteria, or who meet any of the following criteria:

  * Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis.
  * PHOTOSENSITIVITY: Hypersensitivity to sunlight or UVB light of any type; history of Lupus, PMLE, or any disease known to be worsened by UV light exposure
  * A history of non-melanoma skin cancer may be acceptable, and in this situation, the patient will be carefully evaluated.
  * Poorly controlled medical conditions of any kind.
  * Any medical condition that, in the opinion of the Investigator, would jeopardize the health or well being of the patient during the course of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is genomic analysis of lesional skin biopsies, in a time course experiment,by microarray and RT-PCR. | End of study

SECONDARY OUTCOMES:
cell counts of leukocytes populations in skin biopsies including (but not limited to) myeloid dendritic cells (CD11c and CD1c/BDCA-1), plasmacytoid dendritic cells (BDCA-2/CD123), macrophages (CD163), and T cells (CD3, CD4, CD8, Foxp3, RORγ). | End of study
Effects of NB-UVB on NL skin will be determined by comparison of microarray analysis of NL skin biopsies throughout treatment. | End of study
To determine if there is a set of genes that can predict response, expressed in circulating PBMCs, we will perform microarray on baseline PBMCs, and compare the gene sets for responders and non-responders (discriminant analysis). | End of study
To evaluate if treatment causes an altered ratio of Th17:Tregs in the circulation and skin, we will perform intracellular cytokine staining by flow cytometry on peripheral blood and from the shave biopsy. | Before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lowes, MD, PhD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States